CLINICAL TRIAL: NCT02782520
Title: Comparison of the Effects of an Hypertonic Solution With Ringer Lactate on Right Ventricular Function Following Cardiac Surgery
Acronym: SUCCESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38RC15.214
Record Dates: First submitted 2016-04-29; First posted 2016-05-25 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2017-11

CONDITIONS: Right Ventricular Impaired Function; Hypovolemia
Keywords: Cardiopulmonary bypass; Swan Ganz; Fluid expansion; hypertonic saline solution
MeSH Terms: conditions — Hypovolemia | interventions — Ringer's Lactate; Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ringer Lactate (Active Comparator): Ringer Lactate group
  Interventions: Drug: Ringer Lactate (10ml/kg) fluid expansion
- Hypertonic saline (Experimental): Hypertonic saline group
  Interventions: Drug: Hypertonic saline (3ml/kg) fluid expansion

INTERVENTIONS:
Drug: Ringer Lactate (10ml/kg) fluid expansion
  Arms: Ringer Lactate
Drug: Hypertonic saline (3ml/kg) fluid expansion
  Arms: Hypertonic saline

SUMMARY:
This study is a phase III, randomized, controled, parallel groups, single blinded, clinical trial that aims at comparing the improvement of right ventricular function after administration of a hypertonic solution versus Ringer Lactate following cardiac surgery.

Adults patients admitted to Grenoble University Hospital for elective cardiac surgery under cardiopulmonary bypass, in sinus rhythm and with Swan Ganz monitoring will be included.

Patients needing fluid expansion in the first three hours after surgery will be randomized in two groups : one receiving Ringer Lactate (10 mL/kg), the other receiving hypertonic saline solution (3 mL/kg).

Right ventricular function measured with Swan Ganz catheter, 30 minutes after fluid expansion will be the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Elective valvular or coronary surgery
* Under cardiopulmonary bypass
* Patient requiring Swan Ganz catheter monitoring
* Patient in sinus rhythm
* Patient requiring post-operative volemic expansion
* Echographic criteria of hypovolemia, without hypervolemia

Exclusion Criteria:

* Pulmonary hypertension (SPAP > 60mmHg)
* No pre-operative sinus rhythm
* Emergency surgery
* Age < 18 years
* Chronic renal failure treated with dialysis
* Severe hypernatremia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Right ventricular ejection fraction change measured by Swan Ganz catheter. | after 30 minutes perfusion ( fluid expansion)

SECONDARY OUTCOMES:
Left ventricular contractility | at 30, 60 minutes and 3, 6 and 18 hours after perfusion
Systolic volume change | at 30, 60 minutes and 3, 6 and 18 hours after perfusion
Cardiac output evolution. | at 30, 60 minutes and 3, 6 and 18 hours after perfusion
Tricuspid annular plane systolic excursion assessment | One hour before and after perfusion
Continuous cardiac output | at 30, 60 minutes and 3, 6 and 18 hours after perfusion
Blood volume efficiency | One hour before and 30, 60 minutes and 3, 6 and 18 hours after perfusion
  Blood volume efficiency included : Right systolic and diastolic ventricular volumes, measured by swan ganz catheter, central veinous pressure
Plasmatic volume monitoring | One hour before and , 1, 6 and 18 hours after perfusion
  Plasmatic volume augmentation assessed by hemoglobin decrease
Natremia level | at 1, 6 and 18 hours after perfusion
Veinous oxygen saturation | at 30, 60 minutes and 3, 6 and 18 hours after perfusion
Mean arterial pressure assessment. | at 30, 60 minutes and 3, 6 and 18 hours after perfusion
Lactatemia level | at 1, 6 and 18 hours after perfusion
Acid base balance assessment. | at 1, 6 and 18 hours after perfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Reanimation Cardiovasculaire Et Thoracique, La Tronche, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaul TK, Fields BL. Postoperative acute refractory right ventricular failure: incidence, pathogenesis, management and prognosis. Cardiovasc Surg. 2000 Jan;8(1):1-9. doi: 10.1016/s0967-2109(99)00089-7. PMID 10661697
- [Background] Gavazzi A, Berzuini C, Campana C, Inserra C, Ponzetta M, Sebastiani R, Ghio S, Recusani F. Value of right ventricular ejection fraction in predicting short-term prognosis of patients with severe chronic heart failure. J Heart Lung Transplant. 1997 Jul;16(7):774-85. PMID 9257260
- [Background] Christakis GT, Fremes SE, Weisel RD, Ivanov J, Madonik MM, Seawright SJ, McLaughlin PR. Right ventricular dysfunction following cold potassium cardioplegia. J Thorac Cardiovasc Surg. 1985 Aug;90(2):243-50. PMID 3875003
- [Background] Durand M, Chavanon O, Tessier Y, Casez M, Gardellin M, Blin D, Girardet P. Right ventricular function after coronary surgery with or without bypass. J Card Surg. 2006 Jan-Feb;21(1):11-6. doi: 10.1111/j.1540-8191.2006.00161.x. PMID 16426341
- [Background] Mouren S, Delayance S, Mion G, Souktani R, Fellahi JL, Arthaud M, Baron JF, Viars P. Mechanisms of increased myocardial contractility with hypertonic saline solutions in isolated blood-perfused rabbit hearts. Anesth Analg. 1995 Oct;81(4):777-82. doi: 10.1097/00000539-199510000-00021. PMID 7574010
- [Background] Ueti OM, Camargo EE, Ueti Ade A, de Lima-Filho EC, Nogueira EA. Assessment of right ventricular function with Doppler echocardiographic indices derived from tricuspid annular motion: comparison with radionuclide angiography. Heart. 2002 Sep;88(3):244-8. doi: 10.1136/heart.88.3.244. PMID 12181215
- [Background] Hammarstrom E, Wranne B, Pinto FJ, Puryear J, Popp RL. Tricuspid annular motion. J Am Soc Echocardiogr. 1991 Mar-Apr;4(2):131-9. doi: 10.1016/s0894-7317(14)80524-5. PMID 2036225
- [Background] Romano SM. Cardiac cycle efficiency: a new parameter able to fully evaluate the dynamic interplay of the cardiovascular system. Int J Cardiol. 2012 Mar 8;155(2):326-7. doi: 10.1016/j.ijcard.2011.12.008. Epub 2011 Dec 22. No abstract available. PMID 22197117
- [Background] Scolletta S, Bodson L, Donadello K, Taccone FS, Devigili A, Vincent JL, De Backer D. Assessment of left ventricular function by pulse wave analysis in critically ill patients. Intensive Care Med. 2013 Jun;39(6):1025-33. doi: 10.1007/s00134-013-2861-8. Epub 2013 Mar 9. PMID 23474659